CLINICAL TRIAL: NCT02017834
Title: Does the Harmonic Scalpel Reduce Operating Time and Blood Loss in Patients Undergoing Major Surgery for Oral Cavity Squamous Cell Carcinoma? A Prospective, Randomized Trial.
Brief Title: Does the Harmonic Scalpel Reduce Blood Loss and OR Time in Major Head and Neck Cancer Surgery Undergoing Major Surgery for Oral Cavity Squamous Cell Carcinoma?
Acronym: HS2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Joseph C. Dort, Ohlson Professor of Head & Neck Surgery, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UCENT005
Record Dates: First submitted 2012-01-31; First posted 2013-12-23 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2013-12

CONDITIONS: Oral Cavity Squamous Cell Carcinoma, Treated With Surgery
Keywords: oral cavity squamous cell carcinoma; head and neck cancer; oral cancer
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms; Mouth Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- harmonic scalpel (Experimental)
  Interventions: Procedure: surgical resection
- standard technique (Active Comparator)
  Interventions: Procedure: surgical resection

INTERVENTIONS:
Procedure: surgical resection — neck dissection and tumour resection will be performed either with or without the harmonic scalpel as an adjunct.
  Other Names: Harmonic Focus handpiece

SUMMARY:
The harmonic scalpel is a tool that may reduce operative blood loss. Some studies also indicate it may result in faster surgery. A recently published randomized study from our group shows the harmonic scalpel reduces blood loss in neck dissection but it did not offer any reduction in OR time. The present study investigates the utility of the harmonic scalpel in resections involving removal of oral cavity tissues as well as the neck. Oral cavity resections are especially prone to blood loss and we believe the harmonic scalpel will confer benefits in this type of surgery, potentially reducing the need for blood transfusion.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* oral cavity scc
* primary surgery including either uni or bilateral neck dissection (levels I-IV)

Exclusion Criteria:

* previous treatment for head and neck cancer
* unable or unwilling to give informed consent
* history of bleeding disorder
* other contraindications to surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-02; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
blood loss | intraoperative

SECONDARY OUTCOMES:
operating time | intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Dort, MD, Principal Investigator — University of Calgary
Locations (1):
- Foothills Hospital, Calgary, Alberta, Canada

REFERENCES:
- [Derived] Fritz DK, Matthews TW, Chandarana SP, Nakoneshny SC, Dort JC. Harmonic scalpel impact on blood loss and operating time in major head and neck surgery: a randomized clinical trial. J Otolaryngol Head Neck Surg. 2016 Nov 8;45(1):58. doi: 10.1186/s40463-016-0173-z. PMID 27821144